CLINICAL TRIAL: NCT05875896
Title: Investigation of the Functional Status After Wrist Arthrodesis (Medartis Aptus Model) in Patients With Rheumatoid Arthritis Compared to Patients With Post-traumatic Wrist Destruction
Brief Title: Study of Wrist Fusions With the Medartis Aptus Arthrodesis Plate
Acronym: STIF
Status: Completed | Type: Observational
Sponsor: Waldfriede Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BB040/23
Record Dates: First submitted 2023-05-02; First posted 2023-05-25 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Wrist Arthritis; Wrist Osteoarthritis
Keywords: Wrist fusion,Arthrodesis,Rheumatoid Arthritis,Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis wrist destruction: Patients with rheumatoid arthritis who received an APTUS wrist fusion system after 01.01.2014
  Interventions: Procedure: Total wrist fusion
- Osteoarthritis wrist destruction: Patients with post-traumatic wrist osteoarthritis who received an APTUS wrist fusion system after 01.01.2014
  Interventions: Procedure: Total wrist fusion

INTERVENTIONS:
Procedure: Total wrist fusion — Observation after implantation of Medartis Aptus Wrist Arthrodesis Plate

SUMMARY:
The primary working hypothesis of this study is whether wrist arthrodesis leads to an improvement in functional status in both rheumatoid arthritis and post-traumatic osteoarthritis. Functional status will be measured by Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire no earlier than 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-90
* Wrist fusion took place between 2014 and 2022 using Aptus 2.5 TriLock Total Wrist Fusion Plate, Medartis at Hospital Waldfriede
* rheumatoid Arthritis
* post-traumatic osteoarthritis patterns: 1. scapholunate advanced collapse (SLAC) or 2. scaphoid nonunion advanced collapse (SNAC)

Exclusion Criteria:

* post surgery bone fracture of the same limb
* Pregnancy, lactation
* active malignant tumor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have either suffered wrist destruction due to rheumatiod arthritis inflammation, or individuals who have received wrist fusion due to post-traumatic osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand questionnaire (DASH) | all patients who underwent surgery between 2014 to 2022
  Disabilities as measured by the DASH scale; No Difficulty (1), Mild Difficulty (2), Moderate Difficulty (3), Severe Difficulty (4), Unable (5)

SECONDARY OUTCOMES:
Postoperative complications | all patients who underwent surgery between 2014 to 2022
  Number of Participants with impaired wound healing, Re-surgery, Material loosening
Function | all patients who underwent surgery between 2014 to 2022
  Grip force of the hand in Kg
Functional assessment: Goniometry | all patients who underwent surgery between 2014 to 2022
  ROM of each joint of the hand with a goniometer.
Visual analogue scale (VAS) Pain | all patients who underwent surgery between 2014 to 2022
  From 0mm (no pain) to 100mm (maximum pain imaginable)
Short-Form 36 (SF-36) | all patients who underwent surgery between 2014 to 2022
  Scored review of health questionnaire SF36: minimum value = 0 ; maximum value = 100

CONTACTS AND LOCATIONS:
Overall Officials: Lautenbach Martin, MD, Study Chair — Hospital Waldfriede, Argentinische Allee 40, 14163 Berlin; Markus Bock, MD, Principal Investigator — Hospital Waldfriede, Argentinische Allee 40, 14163 Berlin
Locations (1):
- Waldfriede Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided